CLINICAL TRIAL: NCT04711668
Title: The Effect of Introperative Ketamine and Lidocaine Infusion on Postoperative Opioid Consumption in Posterior Spinal Fusion Surgery - Double-Blind Randomized Controlled Study
Brief Title: Effect of Introperative Ketamine and Lidocaine Infusion on Postoperative Opioid Consumption in Posterior Spinal Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vedat Öztürk, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/308
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Spine Fusion; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Ketamin (Experimental): 0.5 mg / kg i.v. ketamine bolus at induction and 0.25 mg / kg / hr i.v. ketamine infusion intraoperatively
  Interventions: Drug: Ketamine
- Group Lidokain (Experimental): 1.5 mg / kg i.v. lidocaine bolus at induction and 1.5 mg / kg / hr i.v. lidocaine infusion intraoperatively
  Interventions: Drug: Lidocain
- Group Placebo (Placebo Comparator): i.v. saline (in the same volume and duration like group ketamine/lidokain)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — intraoperative ketamine bolus and infusion
  Arms: Group Ketamin
Drug: Lidocain — intraoperative lidocain bolus and infusion
  Arms: Group Lidokain
Drug: Saline — intraoperative saline bolus and infusion
  Arms: Group Placebo

SUMMARY:
Objective: The primary aim of this study was to investigate the effect of ketamine and lidocaine on postoperative opioid consumption in posterior spinal fusion surgery.

Materials and Methods: Ethics committee approval was received from our faculty. Seventy-five cases between the ages of 18-65, who have an ASA (American Society of Anesthesiologists) risk classification I-II-III in the preanesthetic evaluation, planned to be operated by the Neurosurgery clinic for lumbar posterior spinal fusion surgery under elective conditions have been included in the study after the informed volunteer consent form was read and approved.

The patients were randomly divided into 3 groups using the closed envelope method. The ketamine group (Group K) (n = 25), the lidocaine group (Group L) (n = 25) and the placebo group (Group P) (n = 25). Propofol, rocuronium and fentanyl i.v. done. In group K, 0.5 mg / kg i.v. ketamine bolus and 0.25 mg / kg / hr i.v. ketamine infusion was administered. In group L, 1.5 mg / kg i.v. lidocaine bolus and 1.5 mg / kg / hr i.v. lidocaine infusion was administered. In group P, i.v. saline (in the same volume and duration) was applied. Maintenance of anesthesia was provided by propofol and remifentanil infusion. The propofol and remifentanil doses were adjusted according to the BIS monitoring and the increase or decrease in basal blood pressure and heart rate values of 20% or more. The BIS value was kept between 40-60. At the end of surgery, infusions were closed. After extubation, the patients were taken to the recovery room. Patient controlled analgesia (PCA) prepared with fentanyl was applied to the patients for postoperative analgesia. The PCA device was attached for 24 hours postoperatively.

Postoperative 0-4 hours, 4-8 hours, 8-24 hours and total fentanyl consumption of the patients were evaluated. Pain scores were measured at 1, 2, 4, 8, 12 and 24 hours in the postoperative recovery room. Intraoperative propofol and remifentanil consumption was recorded. Tramadol 1 mg / kg i.v. as rescue analgesia (in patients with VAS pain score of 4 and above) done. Possible side effects due to opioid, ketamine and lidocaine were followed.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65, who have an ASA (American Society of Anesthesiologists) risk classification I-II-III

Exclusion Criteria:

* Previous spinal surgery, Morbid obesity (BMI> 35 kg / m2), Lidocaine, ketamine or opioid allergy. Severe cardiac or pulmonary disease, Liver or kidney dysfunction Poorly controlled hypertension, Substance abuse, Chronic opioid use, Pregnancy, Psychiatric disorder, Cognitive impairment History of stroke, head injury, and intracranial mass or bleeding and patients who did not want to participate in the study were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | postoperative 0-24 hours
  postoperative PCA wit fentanyl

SECONDARY OUTCOMES:
postoperative pain score | postoperative 0-24 hours
  pain score is visual analogue scala

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided